CLINICAL TRIAL: NCT04637282
Title: A Randomized. Multicenter, Double-Blind, Placebo-Controlled Safety, Tolerability, and Efficacy Study of PLX-200 in Participants With Mild-to-Moderate Juvenile Neuronal Ceroid Lipofuscinosis (CLN3) Disease
Brief Title: Safety, Tolerability, and Efficacy of PLX-200 in Patients With CLN3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Polaryx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLX-200-002
Record Dates: First submitted 2020-11-04; First posted 2020-11-19 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Juvenile Neuronal Ceroid Lipofuscinosis
Keywords: CLN3; Batten disease; Children
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses | interventions — Gemfibrozil

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, within-subject, dose-titration design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PLX-200 (Experimental): This is randomized, placebo-controlled comparator study of PLX-200 in patients with CLN3 disease.
  Interventions: Drug: PLX-200
- Placebo (Placebo Comparator): This is randomized comparator study of PLX-200 vs. placebo in a 2:1 ratio in patients with CLN3 disease.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PLX-200 — 15 mg/mL oral solution of experimental drug
  Other Names: Gemfibrozil
  Arms: PLX-200
Drug: Placebo — Taste and color-matched drug-free solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of multiple doses of PLX-200 in patients with CLN3 disease.

DETAILED DESCRIPTION:
This is a phase 3, double-blind, placebo-controlled, dose-titration study to evaluate escalating weight-based dose levels of PLX-200, provided as a solution that contains 15 mg/mL PLX-200 and administered orally using a syringe, as needed, twice daily (BID), 30 minutes before breakfast and dinner. Participants will enter the Titration Period, during which the starting dose of PLX-200 or placebo will be based on patient weight. Each patient's dose will be titrated upward on a weekly basis during the Titration Period, until he or she reaches a maximally tolerated dose (MTD) or the Week 5 dose for their weight category. The patient will then enter the Maintenance Period at the final Titration Period dose for a maximum of 60 weeks. Safety, efficacy, and pharmacokinetics will be assessed periodically. Thereafter, all patients will have the opportunity to receive active treatment in an Open-Label Extension (OLE) for an additional 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants between the ages of 6 and 18 years of age. Any deviations from this age range must be approved by the Medical Monitor and Sponsor prior to entry into study.
2. Has a diagnosis of "classic" CLN3 disease as determined by age of symptom onset (i.e., 4 to 7 years) and genetic analysis for a defect in the CLN3 (battenin) transmembrane gene at study entry. If no genotype information is available, blood will be collected for the CLN3 gene analysis at the Screening visit.
3. Participant must have mild-to-moderate CLN3 disease documented by a total in the 3-domain score of 5 to 7 for the aggregate of the motor, language, and vision domains of the Hamburg Scale and a score of at least 2 in 2 of these 3 domains.
4. Participant must be able to independently walk for a distance of at least 20 feet (6 meters).
5. Participant must be able to tolerate swallowing oral medication.
6. Participants who are of childbearing potential (i.e., have begun menstruation) must have a negative serum pregnancy test at Baseline before receiving PLX-200. Nursing mothers are excluded from participation in this study.
7. Participants' parents/guardians must agree to comply in good faith with the conditions of the study, including attending all required baseline and follow-up assessments.
8. Participant parents and legal guardians must sign the informed consent form, and participants will provide assent, depending on local regulations and developmental status.

Exclusion Criteria:

1. Participant has asymptomatic CLN3 disease, defined as no evidence of neurological signs or symptoms attributed to CLN3 disease such as seizures, ataxia, language delay, or other developmental delays. Similarly, outliers who progress much more slowly or quickly compared to the rest of the study population will be excluded from study at the discretion of the PI in consultation with the Medical Monitor (e.g., c.1A > C start codon mutation).
2. Participant has clinically documented generalized motor status epilepticus within 4 weeks of the Baseline visit (treatment may be postponed after discussion with the Medical Monitor until seizures are adequately controlled).
3. Participant has another inherited neurologic disease in addition to CLN3 disease.
4. Participant has another neurological illness that may cause cognitive or motor decline.
5. Participants with enteral feeding with NG tubing and any difficulty in oral administration and/or absorption of study drug will be excluded.
6. Participant requires ventilation support, except for noninvasive support at night (e.g., Continuous Positive Airway Pressure [CPAP], Bilevel Positive Airway Pressure [BiPAP]).
7. Participant has moderate or severe hepatic dysfunction defined as alanine aminotransferase, aspartate aminotransferase, or total bilirubin >3x upper limit of normal (ULN) except for participants with Gilbert syndrome. Participant has primary biliary cirrhosis.
8. Participant has anemia (defined as hemoglobin <10 g/dL or hematocrit <30%).
9. Participant has a baseline serum creatinine >2 mg/dL.
10. Participant has gallbladder disease (e.g., cholelithiasis or cholecystitis).
11. Participant has hypersensitivity to gemfibrozil.
12. Participant is using or requires treatment with 1. HMG-CoA reductase inhibitors, 2. repaglinide (Prandin®), 3. dasabuvir (Exviera®), 4. selexipag (Uptravi®), or 5. pioglitazone (Actos®).
13. Since the participant may take anticoagulants, increased frequency of INR monitoring is essential to avoid potential toxic effects with concurrent PLX-200 and anticoagulants (in particular with warfarin).
14. Participant has a medical condition or personal circumstance that, in the opinion of the Investigator, might compromise the participant's or parent/guardian's ability to comply with the protocol requirements, or compromise the participant's wellbeing, safety, or the interpretability of the study data.
15. Participant has received any investigational product or medical device within 30 days of the Baseline visit that, in the Investigator's judgment, would make the participant ineligible or confound results. All subjects who have had an investigational product or products in the form of stem cell or gene therapy are excluded, regardless of when the therapy had been initiated and/or discontinued.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of PLX-200 in CLN3 as assessed by the change in the motor score of the Hamburg Rating Scale compared with that of the Placebo group | 60 weeks
  The change from baseline in the motor score of the Hamburg Rating Scale at Week 60 of maintenance therapy in participants treated with PLX-200 compared with that of Placebo group. Baseline is defined as the motor score of the Hamburg Rating Scale assessment prior to starting drug or Placebo group in the Titration Period. The Hamburg Rating Scale records a rating of 0 - 3 in four domains: motor skills, vision, language, and seizures, all from 0 - 3 which is worse to normal, respectively, with a minimum (worse) score of 0 to a maximum (normal) score of 12.
Number of patients with treatment-related adverse events, as assessed by CTCAE v5.0, abnormal laboratory results, and abnormal cardiovascular and/or abdominal findings. | 96 weeks
  The aggregate of clinical chemistries, hematology, urinalysis, electrocardiogram readings, abdominal ultrasound findings, and tabulation of the number and severity of adverse events will be compared with baseline values throughout the study to evaluate the safety and tolerability of PLX-200 at escalating oral doses in children with CLN3 disease.

SECONDARY OUTCOMES:
Efficacy of PLX in each of the domains of the Hamburg Scale | 24, 48, 60, 72 and 96 weeks
  Changes in the Baseline score of each of the 4 domains of the Hamburg Rating Scale (motor, language, visual, and seizures) at 24, 48, 60 (except motor score), 72, and 96 weeks of maintenance therapy in those treated with PLX-200 compared with those treated with Placebo. The Hamburg rating per domain is 0 - 3 with 3 representing worse outcomes.
Assessment of the overall decline status in subjects treated with PLX-200 compared with the placebo group | 60 and 96 weeks
  The overall decline status (Yes/No) at Maintenance Weeks 60 and 96 in subjects treated with PLX-200 compared to those treated with Placebo. A subject will be considered to have an overall decline if either (i) a decrease from baseline in any of the 4 domains (motor, language, visual, seizure) of the Hamburg rating scale is observed or (ii) the assessment is missing at the visit for any reason. The Hamburg rating per domain is 0 - 3 with 3 representing worse outcomes.
Evaluation of the baseline motor score decline between PLX-200 and placebo | 60 and 96 weeks
  The Motor Score decline status (Yes/No) at Maintenance Weeks 60 and 96 in subjects treated with PLX-200 compared to those treated with Placebo using two alternative definitions. In Definition 1, a subject will be considered to have declined (i.e. worsened) if at least a one-point decrease from baseline in the motor score of the Hamburg scale is observed or if the visit is missing for any reason. In Definition 2, subjects with at least a 2-point decrease or if the visit is missing will be considered to have declined.
Assessment of changes in the baseline Clinical Impression of symptom severity between PLX-200 and Placebo groups | 24, 48, 60, 72, and 96 weeks
  Changes from baseline in the Clinical Global Impression of symptom severity to 24, 48, 60, 72, and 96 weeks of maintenance therapy in those treated with PLX-200 compared with those treated with Placebo. The CGI severity scale (CGI-S) rates illness severity and the CGI-Improvement (CGI-I) which both rate on a scale of 1 - 7 which relates to improved/very much improved to worse disease.
Assessment of changes in the baseline Pediatric Balance Scale between PLX-200 and Placebo groups | 24, 48, 60, 72, and 96 weeks
  Change in the Pediatric Balance Scale (modified Berg Balance Scale) score from Baseline to 24, 48, 60, 72, and 96 weeks of maintenance therapy in those treated with PLX-200 compared with those treated with Placebo. The scale is age, weight, height, and gender specific but across all groups, the higher score between 0 - 4 represents better outcomes than 0 which is worse outcome.
Assessment of changes in the baseline Montreal Assessment Cognitive Scale between PLX-200 and Placebo groups | 24, 48, 60, 72, and 96 weeks
  Change in the Montreal Cognitive Assessment (MoCA) score from Baseline to 24, 48, 60, 72, and 96 weeks of maintenance therapy in those treated with PLX-200 compared with those treated with Placebo. The MoCA cutoff score of 26 differentiates youth with and without cognitive impairment with the lower score being considered increased cognitive impairment.
Assessment of changes in the baseline Vineland Behavior Scale between PLX-200 and Placebo groups | 24, 48, 60, 72, and 96 weeks
  Change in the Vineland Behavior Scale from Baseline to 24, 48, 60, 72, and 96 weeks of maintenance therapy in those treated with PLX-200 compared with those treated with Placebo. The Vineland Scale captures changes in intellectual and developmental disabilities. To date, there are no normal values determined for the Vineland Behavior Scale but the higher the score suggests greater capabilities.
Assessment of changes in the baseline walking ability of the patient between PLX-200 and Placebo groups | 24, 48, 60, 72, and 96 weeks
  Change in walking ability (6-minute walk test; 6MWT) from Baseline to weeks 24, 48, 60, 72, and 96 weeks of maintenance therapy in those treated with PLX-200 compared with those treated with Placebo. The 6MWT normal range is highly specific to the patient. Thus, all tests will be compared to the Baseline value during the Screening Phase.
PLX-200 pharmacokinetics (PK) will be evaluated through periodic blood draws during the trial. PLX-200 levels will be determined to estimate area under the curve, maximal concentration, time to maximal concentration, half-life, and dosing interval | 96 weeks
  To evaluate PLX-200 plasma concentrations in blood collected from participants during the Titration and Maintenance Periods for PK analyses, namely Cmax (maximal PLX-200 concentration) and Tmax (time to Cmax), elimination half-life (t1/2), area under the plasma concentration-time curve (AUC), and the dosing interval.

IPD SHARING:
Plan to Share IPD: No
None planned.